CLINICAL TRIAL: NCT01959724
Title: Macular Detachment Associated With Intrachoroidal Cavitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Associate professor of Ophthalmology, Kyorin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kyorineye012; Kyorineye12 (Other: Kyorin Eye Center)
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Macular Detachment; Macular Retinoschisis; Intrachoroidal Cavitation
Keywords: Macular detachment; Macular retinoschisis; Vitrectomy
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitrectomy (Other): Vitreous surgery to treat macular detachment
  Interventions: Other: Vitrectomy

INTERVENTIONS:
Other: Vitrectomy

SUMMARY:
Evaluation of clinical characteristics and surgical outcome for macular detachment associated with peripapillary intrachoroidal cavitation with or without pathologic myopia.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with macular detachment or macular retinoschisis

Exclusion Criteria:

* Optic pit maculopathy, vitreomacular traction syndrome

Ages: 10 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-04; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Visual acuity | one year
  The numbers of the patients with visual recovery after surgical intervention

SECONDARY OUTCOMES:
Optical coherence tomography | one year
  Anatomical improvement detected with optical coherence tomography after surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Kyorin Eye Center
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan